CLINICAL TRIAL: NCT05146388
Title: Leveraging the EHR to Promote Pharmacy Adoption of Dosing Best Practices and Reduce Parent Errors in Administering Pediatric Liquid Medications: A Health Literacy-Informed Approach
Brief Title: Working With Doctors and Pharmacists to Help Parents Give Children's Liquid Medicines Safely
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 21-00972
Record Dates: First submitted 2021-11-23; First posted 2021-12-06 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Medication Dosing Error
Keywords: Electronic Prescriptions (e-Rx); Pharmacy Dispensing Practices

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single (Outcomes Assessor) Two raters will independently assess dosing errors. Raters will be kept blinded to each other's estimated dose volumes and dosing error assessment in order to minimize bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-Implementation - Usual Care (No Intervention): In pre-implementation phase, patient e-Rxs will be generated by the EHR in the usual fashion.
- Post-Implementation - EHR-Based Approach (Experimental)
  Interventions: Other: EHR-Based Approach

INTERVENTIONS:
Other: EHR-Based Approach — The intervention will be built directly into the EHR. E-prescriptions will be generated with pharmacy instructions for all prescription medications. The intervention will impart: 1) inclusion with e-Rx request for pharmacy to keep metric-only (mL-only) dosing on Rx label and 2) inclusion of guidance on the e-Rx requesting that the pharmacy give an optimal tool based on an algorithm. Algorithm for dosing tool recommendation: 1) for a prescribed dose of <= 1mL, optimal tool is 1 mL syringe, 2) for >1 mL to 5 mL, use a 5 mL syringe, 3) for >5mL to 10mL, use 10 mL syringe.
  Arms: Post-Implementation - EHR-Based Approach

SUMMARY:
The study objective is to assess the impact of an automated electronic health record (EHR)-based intervention that leverages e-prescriptions to support pharmacist adherence to recommended dispensing practices, with the goal of reducing parent dosing errors.

Specifically, the study aims are to: 1) Examine the efficacy of the EHR-based intervention in improving pharmacy dispensing practices, including a) adherence to mL-only dosing and b) provision of optimal dosing tools; 2) Examine the efficacy of the EHR-based intervention in reducing parent dosing errors. The study will also explore whether implementation of the EHR-based intervention will reduce disparities in dosing errors by parent health literacy and LEP, and explore the efficacy of the EHR-based intervention in reducing ADEs.

A pre-/post-implementation study will be performed with English- and Spanish-speaking parents of children prescribed oral liquid medications in the pediatric emergency room, outpatient general pediatric clinic, and pediatric subspecialty clinics of 2 New York City hospital systems (NYU Langone Health - Brooklyn and NYC Health+Hospitals - Bellevue Hospital). Prior to implementation, e-Rx's will be generated by the EHR in the usual fashion; after implementation, e-Rx's will be generated by the EHR with instructions to the dispensing pharmacy to: 1) keep the dosing instructions in mL-only, and 2) dispense a specific dosing tool based on the amount prescribed.

The proposed project is consistent with a growing national focus on promoting the adoption of evidence-based strategies to improve disease management that address the needs of those with low health literacy and LEP from groups like the Joint Commission and the AHRQ.

ELIGIBILITY:
Inclusion Criteria:

Caregiver/Child

1. English or Spanish-speaking
2. Parent or legal guardian of a child prescribed a liquid medicine in the NYU Langone Health - Brooklyn or Bellevue ED, general outpatient pediatric clinic, or specialty care clinics
3. 18 years of age or older
4. Child ≤8y discharged home with a Rx for ≥1 daily liquid medication dose ≤10mL, for use as a chronic or short course (≤14 days) medication
5. Primary person who will administer child's medications
6. Access to a smartphone that can take photos and send/receive text messages
7. Willingness and ability to participate

Pharmacy staff

1. Works at a pharmacy that dispensed index medicine to one of our study participants.

Exclusion Criteria:

Caregiver/Child

1. Does not have a working phone number
2. Not able to return for in-person follow-up visit
3. Was told to stop medication by provider after doctor/ED visit
4. Parent no longer having index medication bottle
5. Uncorrected hearing impairment
6. Self-reported poor visual acuity

Pharmacy staff

1. Staff with no responsibility in determining unit of measure to include on Rx's or type/capacity of the dosing tool to dispense for pediatric oral liquid medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-04-21 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Caregiver Dosing Error | Within 8 weeks of index visit (Visit 2)
  Dosing error will be defined as >20% deviation from the prescribed dose
Caregiver Large Dosing Error | Within 8 weeks of index visit (Visit 2)
  Large dosing error will be defined as >40% deviation from the prescribed dose
Pharmacy Use of mL-only on Rx Label | Within 4 weeks of index visit (Visit 1)
Pharmacy Provision of Optimal Dosing Tool | Within 4 weeks of index visit (Visit 1)

CONTACTS AND LOCATIONS:
Overall Officials: H. Shonna Yin, MD, MS, Principal Investigator — NYU Langone Health
Locations (3):
- United States (3):
  - NYU Langone Health - Brooklyn, Brooklyn, New York
  - Sunset Park Family Health Center at NYU Langone, Brooklyn, New York
  - NYC Health + Hospitals / Bellevue, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to Hsiang.Yin@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.